CLINICAL TRIAL: NCT07236294
Title: Material and Clinical Assessment of 3D-printed vs. Milled Occlusal Splints: A Study on Performance and Durability in Dental Applications
Brief Title: 3D Printed vs. Milled Occlusal Splints in Dentistry
Acronym: Splints
Status: Not yet recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-17704
Record Dates: First submitted 2025-07-22; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2024-11

CONDITIONS: Wear Comfort; Retention; Stability
Keywords: 3D printed splints; Milled splints; Prospective clinical randomized crossover study; Retention; Stability; comfort

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This crossover study aims to evaluate the wear comfort, retention, and stability of 3D-printed and milled occlusal splints in healthy subjects.

The main question it aims to answer is:

Research questions

- How do healthy subjects experience the wear comfort, fitting, retention and stability of a printed and milled occlusal splint? and how do clinicians experience the fitting, retention and stability of the splints?

By systematically assessing self-reported outcomes, this research seeks to contribute valuable insights into the practical applications of both technologies. The findings may not only enhance our understanding of patient preferences but also guide future developments in the design and manufacturing of occlusal splints, ultimately improving patient care in dental practice.

DETAILED DESCRIPTION:
The main study parameter is to assess the participant self-reported findings regarding the comfort, retention, stability and fit of the milled and printed splint and in addition to the hygiene and discoloration of the splint over time.

ELIGIBILITY:
Inclusion Criteria:

* Subjects being healthy (ASA <IV)
* Subjects with healthy, complete dentitions (except for extractions of wisdom teeth, or tooth extractions for the purpose of orthodontic treatment in the past)
* Subjects willing and able to participate in the study
* Subjects willing to provide written informed consent for their participation in the study

Exclusion Criteria:

* Subjects with dental issues other than the inclusion criteria
* Subjects with a history of autoimmune disorder
* Subjects with known allergies to acrylic materials
* Subjects with severe allergies manifested by a history of anaphylaxis or those with severe, chronic allergies (e.g., asthma) and subjects with an active infection of any kind at the time of enrollment
* Subjects who are pregnant or lactating
* Subjects enrolled in another investigational clinical trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population for this prospective clinical randomized crossover trial, will consist of young adult participants aged 18 to 45, which study Dentistry, or are a co-worker or patient at the Dentistry Department of Radboudumc Nijmegen.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Comfort | "From enrollment to the end of treatment at 6 weeks"
  Self reported wear comfort by filling in a questionnaire. This scale measures the comfort of the occlusal splint, where "Very uncomfortable" represents the worst experience (lowest score) and "Very comfortable" represents the best experience (highest score). Minimum Value: Very uncomfortable, Maximum Value: Very comfortable. Higher Scores Mean: Better comfort (more comfort)

SECONDARY OUTCOMES:
Stability | From enrollment to the end of treatment at 6 weeks
  Two dentists will evaluate the splints outside of the mouth using a standardized assessment form (pre-tested) focussing on stability. The splints will then be placed in the mouth of the subject and reassessed based on the same parameter.
  Description: This is a custom-developed 5-point Likert-type scale designed to assess the experience of splint stability. Dentists rate how stable or mobile the occlusal splint feel.
  Scale Values:
  1. = Very unstable / significant movement
  2. = Unstable / some movement
  3. = Neutral / no notable instability or discomfort
  4. = Stable / little to no discomfort
  5. = Very stable / no movement or discomfort at all Score Range: Minimum = 1, Maximum = 5 Higher scores indicate a better outcome (i.e. greater stability and comfort during wear).
  Participants also rate stability on the same way. They rate how stable or mobile the occlusal splint felt during use.
Perceived Retention of Occlusal Splint on Model | From enrollment to end of treatment at six weeks
  This 5-point Likert-type scale measures the perceived retention (fit and tightness) of the splint when seated on the dental model, used to assess passive fit.
  Scale Values:
  1. = Much too loose
  2. = Loose, but acceptable
  3. = Optimal
  4. = Slightly tight, but acceptable
  5. = Too tight Score Range: Minimum = 1, Maximum = 5 A score of 3 ("Optimal") indicates the ideal result, where the occlusal splint has a good fit and retention on the model.
  Scores 1-2 ("Too loose") and 4-5 ("Too tight") indicate deviations from optimal retention, which may be considered suboptimal and might require adjustment.
Perceived Retention of Occlusal Splint During Wear | From enrollment to the end of treatment at six weeks.
  A custom 5-point Likert-type scale measuring how well the occlusal splint stays in place during use, based on patient-reported experience. The scale evaluates whether the retention is too loose or too tight, or within acceptable/optimal limits.
  Scale Values:
  1. = Much too loose
  2. = Loose, but acceptable
  3. = Optimal
  4. = Slightly tight, but acceptable
  5. = Very good Score Range: Minimum = 1, Maximum = 5 Directionality: Higher scores indicate a better outcome (i.e. better retention and patient satisfaction during wear).
Perceived Fit of the Occlusal Splint on the Model and in the Mouth | From enrollment to end of the treatment at six weeks.
  This 5-point Likert-type scale evaluates the fit of the occlusal splint both on the dental model and in the patient's mouth. It assesses how well the splint is perceived to conform to the desired shape and fit, both passively on the model and during wear.
  Scale Values:
  1. = Very poor
  2. = Poor
  3. = Average
  4. = Good
  5. = Very good Score Range: Minimum = 1, Maximum = 5
  Directionality:
  Higher scores represent better fit (i.e., optimal adaptation and minimal discomfort).
Perceived Fit of the Occlusal Splint on Teeth | From enrollment to end of the treatment at six weeks
  This 5-point Likert-type scale measures how well the patient feels the occlusal splint fits on their teeth. This includes subjective experiences regarding comfort and fit quality.
  Scale Values:
  1. = Very poor fit
  2. = Poor fit
  3. = Average fit
  4. = Good fit
  5. = Very good fit Score Range: Minimum = 1, Maximum = 5
  Directionality:
  Higher scores indicate a better fit (i.e., a more comfortable and effective splint).
Cleanability | From enrollment to the end of treatment at 6 weeks.
  This 5-point Likert-type scale measures how easy or difficult it is for the patient to keep the occlusal splint clean. It evaluates the patient's experience of cleaning the splint and the effort involved in maintaining its cleanliness.
  Scale Values:
  1. = Very difficult to clean
  2. = Difficult to clean
  3. = Neutral
  4. = Easy to clean
  5. = Very easy to clean Score Range: Minimum = 1, Maximum = 5
  Directionality:
  Higher scores indicate that the splint is easier to clean, suggesting better material or design for cleanliness.
Occlusion | From enrollment to the end of treatment at 6 weeks.
  Articulating paper is used to check the occlusion. The contact marks of the paper help identify areas of contact between the splint and natural teeth, and the distribution of these contacts is assessed.
  1. = Very Poor Occlusion. Few or no contacts, or contacts are isolated in a small area, which may create uneven pressure and discomfort.
  2. = Poor Occlusion. A small number of scattered contacts, or large areas without contact. There are visible areas where the occlusion is uneven.
  3. = Neutral Occlusion. Contacts are generally evenly distributed but may be slightly uneven in certain areas. Some contact marks, but no clear high spots or excessive force.
  4. = Good Occlusion Most contacts are evenly distributed. A few areas may show slightly heavier marks but are within an acceptable range comfort and function.
  5. = Very Good Even pressure across the splint, indicating optimal fit. Higher scores (4-5) indicate better occlusion.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Mechelse, drs., Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: Yes
Specific IPD datasets, such as those underlying published results, will be shared. However, this sharing will occur under strict conditions to ensure data security and participant confidentiality. The data will be pseudonymized, using a secure key management system to separate identifiers from research data. Access will require appropriate agreements, ensuring compliance with ethical and legal standards, and will be granted only for research purposes aligning with the study's objectives.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years after the publication of results.
Access Criteria: To ensure confidentiality and compliance, access to IPD will be restricted to authorized personnel involved in the research process, including the Principal Investigator (PI), specific research team members, external collaborators, and regulatory authorities. Access is based on each individual's role and necessity for the research. The PI will have full access to the IPD, pseudonymized data, and supporting documents for data management and reporting. Research team members, such as co-investigators, assistants, and statisticians, will have access to the data necessary for their assigned tasks. Access will be controlled through formal data requests, Data Use Agreements, and secure platforms. Pseudonymization ensures participant confidentiality while enabling the sharing of valuable research data for scientific progress.